CLINICAL TRIAL: NCT00391456
Title: Use of Animal-Assisted Therapy to Decrease Cardiopulmonary Pressures, Neurohormone Levels, and State Anxiety in Patients Hospitalized With Heart Failure
Brief Title: Animal-Assisted Therapy for Hospitalized Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Pet Care Trust (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: #01061809; ISRCTN26749623
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Heart Failure
Keywords: animal-assisted therapy; dog hospital visit; heart failure
MeSH Terms: conditions — Heart Failure | interventions — Animal Assisted Therapy

INTERVENTIONS:
Behavioral: Animal-assisted Therapy

SUMMARY:
Effects of complementary therapies on heart failure, a leading cause of hospitalization, are unknown. Animal-assisted therapy improves physiological and psychosocial variables in healthy and hypertensive subjects.

The purpose of this study was to determine whether a 12-minute hospital visit with a therapy dog improves hemodynamics, lowers neurohormone levels, and decreases state anxiety in patients hospitalized with heart failure.

DETAILED DESCRIPTION:
Context: Effects of complementary therapies on heart failure, a leading cause of hospitalization, are unknown. Animal-assisted therapy improves physiological and psychosocial variables in healthy and hypertensive subjects.

Objectives: To determine whether a 12-minute hospital visit with a therapy dog improves hemodynamics, lowers neurohormone levels, and decreases state anxiety in patients hospitalized with heart failure.

Design, Setting, Participants: A 3-group (volunteer-dog team, volunteer only, and control) randomized repeated-measures experimental design was used in 76 adult patients with advanced heart failure hospitalized between November 2001 and July 2004. Longitudinal analysis was used to model differences among the 3 groups at 3 time points.

Interventions: One group received a 12-minute visit from a volunteer with a therapy dog, another group received a 12-minute visit from a volunteer, and the control group received usual care, at rest. Data were collected at baseline, 8 minutes after the intervention started, and 16 minutes (4 minutes after intervention ended).

Main Outcome Measures: Blood pressure, heart rate, pulmonary artery pressure, pulmonary capillary wedge pressure, right atrial pressure, cardiac index, systemic vascular resistance, plasma levels of epinephrine and norepinephrine, and state anxiety.

Results: Compared with the control group, patients visited by a volunteer-dog team showed significantly greater decreases in pulmonary artery pressure during (5.34, P = .003) and after (5.78, P = .001) the intervention, pulmonary capillary wedge pressure during (3.09, P = .02) and after (4.31, P = .002) the intervention, and epinephrine (17.54, P = .04) and norepinephrine (240.14, P = .02) levels during the intervention. After the intervention, patients visited by the volunteer-dog team showed the greatest decrease in state anxiety over patients visited by a volunteer only (6.65, P = .003) and the control group (9.13, P < .0001).

Conclusions: Animal-assisted therapy improves cardiopulmonary pressures, neurohormone levels, and anxiety in patients hospitalized with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of heart failure requiring medical management with an indwelling pulmonary artery catheter
* age between 18 and 80 years
* ability to read, write, and speak English
* mental status: alert and oriented to person, place, and time
* SVR greater than 1200 dyne · sec · cm-5 at least once within 12 hours from the start of data collection

Exclusion Criteria:

* SVR less than 1200 dyne · sec · cm-5
* allergies to dogs
* immunosuppression, defined as a white blood cell count of less than 4500 cells/mm3
* infection as determined by an elevated white blood cell count exceeding 11,000 cells/mm3
* body temperature greater than 38ºC
* decreased level of consciousness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76
Dates: Start 2001-11; Study Completion 2004-07

PRIMARY OUTCOMES:
Blood pressure
heart rate
pulmonary artery pressure
pulmonary capillary wedge pressure
right atrial pressure
cardiac index
systemic vascular resistance
plasma levels of epinephrine
plasma levels of norepinephrine
state anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Kathie Cole, RN, MSN, Principal Investigator — University of California, Los Angeles; Anna Gawlinski, RN, DNSc, Principal Investigator — UCLA Medical Center & School of Nursing
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

REFERENCES:
- [Result] Cole K, Gawlinski A, Steers N. Animal assisted therapy decreases hemodynamics, plasma epinephrine and state anxiety in hospitalized heart failure patients. Circulation 112(17 Supplement II):527, 2005.